CLINICAL TRIAL: NCT07224646
Title: Whole-Body Photobiomodulation Use in Professional Soccer Players During a State Championship
Acronym: WBPBM-PSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Italo Amaral de Oliveira, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 84660524.7.0000.5504
Record Dates: First submitted 2025-09-04; First posted 2025-11-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Athletic Performance; Muscle Fatigue; Muscle Strength; Sports
Keywords: Phototherapy; Laser therapy; Muscle fatigue; Muscle damage; Soccer
MeSH Terms: interventions — phytobacteriomycin

STUDY DESIGN:
Intervention Model Description: Model Description:
  Participants are randomly assigned to two parallel groups: an Active Photobiomodulation (PBM) group and a Sham PBM group. Both groups undergo the same training schedule and assessment timeline, but only the active group receives therapeutic light exposure. There is no crossover between groups throughout the 8-week intervention period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-masked trial. Participants wear protective eyewear; the sham device is physically identical and runs the same schedule, fan noise, and indicator covers, but emits no therapeutic light. Operators who run sessions are distinct from outcomes assessors; participants and assessors are unaware of group assignment. Scheduling and room procedures minimize cross-talk between teams. Randomization and assignment are concealed using sealed, opaque envelopes prepared by an independent researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active PBM (Experimental): Whole-body PBM delivered with a Joovv Elite System (6 LED panels; 660±10 nm red and 850±10 nm near-infrared; total panel area ≈12,193 cm²). Athlete stands ~20 cm from panels, wearing eye protection. Two exposures per session: 450 s anterior + 450 s posterior (total 15 min). Measured average irradiance ≈81.62 mW/cm² and energy density per region ≈25.71 J/cm² at 20 cm. Two sessions/week on non-consecutive days for 8 weeks, after routine training.
  Interventions: Radiation: Whole-Body Photobiomodulation (PBM) (Active PBM)
- Sham PBM (Placebo Comparator): Identical setup and schedule, but with therapeutic light disabled (placebo light only). Eye protection and blinding procedures identical to active PBM.
  Interventions: Radiation: Sham PBM

INTERVENTIONS:
Radiation: Whole-Body Photobiomodulation (PBM) (Active PBM) — This intervention consists of whole-body photobiomodulation delivered using a full-body PBM device. Sessions are performed twice weekly on non-consecutive days for 8 weeks, coinciding with the athletes' standard training. The device emits therapeutic light at specified wavelengths and power, targeting the entire body. The protocol is standardized according to prior research, ensuring consistent exposure for all participants in the active arm. The intervention aims to improve muscle performance and recovery while reducing delayed onset muscle soreness (DOMS).
  Arms: Active PBM
Radiation: Sham PBM — Intervention Description (Sham PBM):
  Participants receive a sham photobiomodulation intervention using the same device and schedule, but without emission of therapeutic light. The procedure mimics the active intervention to maintain blinding while allowing comparison of outcomes, including muscle performance, DOMS, and blood markers.
  Arms: Sham PBM

SUMMARY:
This study aims to investigate the effects of whole-body photobiomodulation on professional soccer players during a state championship. The primary question is whether photobiomodulation improves recovery, reduces muscle fatigue, and enhances performance compared to standard training without photobiomodulation.

DETAILED DESCRIPTION:
Detailed Description:

This randomized, controlled clinical trial aims to evaluate the effects of whole-body photobiomodulation (PBM) on recovery and performance in professional soccer players during a state championship.

The intervention will be performed twice weekly on non-consecutive days for 8 weeks, in combination with each athlete's standard training routine. Participants will be allocated to either an active PBM group or a sham PBM group, both following identical procedures to maintain blinding.

Throughout the study, participants will complete scheduled assessments at baseline, during, and after the 8-week period to monitor performance, muscle soreness, and hematological responses. Data will be analyzed using appropriate statistical tests, with a significance level of 5% (two-tailed).

ELIGIBILITY:
Inclusion Criteria:

* Male professional soccer players currently competing in the championship
* Age 18-35 years
* Training frequency ≥5 times per week
* Able to attend all PBM/sham sessions and all assessments during the 8-week intervention
* Signed informed consent

Exclusion Criteria:

* Lower-limb musculoskeletal injury in the last 6 months or currently receiving treatment
* Current use of phototherapy or any other recovery-enhancing modality
* Chronic medical conditions that may affect performance or recovery
* Known sensitivity or contraindication to light-based therapies
* Inability to comply with the intervention or training schedule

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Delayed Onset Muscle Soreness (DOMS) | Baseline (T1), weekly (T2, weeks 1-8), and end of week 8 (T3).
  Pain intensity measured using the Numeric Rating Scale (NRS; 0-10 points; higher scores = worse pain) during a maximal voluntary knee-extension contraction in sitting. Pain location/extent captured with a standardized pain drawing (exploratory). Primary analysis uses NRS.

SECONDARY OUTCOMES:
Knee Extensor Strength (Hand-Held Dynamometry) | Baseline (T1), weekly (T2, weeks 1-8), end of week 8 (T3)
  Peak force of dominant-leg knee extensors measured with a handheld dynamometer in standardized seated position; mean of two MVC attempts used for analysis.
Squat Jump (SJ) Height | Baseline (T1), weekly (T2, weeks 1-8), end of week 8 (T3) Unit: cm
  Vertical jump height (cm) from Squat Jump (SJ) with hands on hips; mean of two trials; flight-time method on contact device.
Countermovement Jump (CMJ) Height | Baseline (T1), weekly (T2, weeks 1-8), end of week 8 (T3)
  Vertical jump height (cm) from Countermovement Jump (CMJ) with hands on hips; mean of two trials; flight-time method on contact device.

CONTACTS AND LOCATIONS:
Overall Officials: Italo A Oliveira, MSc, Principal Investigator — UFSCAR
Locations (1):
- Desportivo Brasil Training Center, Porto Feliz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
At this time, the plan for sharing individual participant data (IPD) has not been determined. Decisions regarding data sharing will be made after study completion, considering participant privacy, ethical approvals, and applicable institutional policies.

REFERENCES:
- [Background] Zagatto AM, Dutra YM, Lira FS, Antunes BM, Faustini JB, Malta ES, Lopes VHF, de Poli RAB, Brisola GMP, Dos Santos GV, Rodrigues FM, Ferraresi C. Full Body Photobiomodulation Therapy to Induce Faster Muscle Recovery in Water Polo Athletes: Preliminary Results. Photobiomodul Photomed Laser Surg. 2020 Dec;38(12):766-772. doi: 10.1089/photob.2020.4803. PMID 33332232
- [Background] Vanin AA, Verhagen E, Barboza SD, Costa LOP, Leal-Junior ECP. Photobiomodulation therapy for the improvement of muscular performance and reduction of muscular fatigue associated with exercise in healthy people: a systematic review and meta-analysis. Lasers Med Sci. 2018 Jan;33(1):181-214. doi: 10.1007/s10103-017-2368-6. Epub 2017 Oct 31. PMID 29090398
- [Background] Van Hooren B, Zolotarjova J. The Difference Between Countermovement and Squat Jump Performances: A Review of Underlying Mechanisms With Practical Applications. J Strength Cond Res. 2017 Jul;31(7):2011-2020. doi: 10.1519/JSC.0000000000001913. PMID 28640774
- [Background] Thong ISK, Jensen MP, Miro J, Tan G. The validity of pain intensity measures: what do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018 Jan 26;18(1):99-107. doi: 10.1515/sjpain-2018-0012. PMID 29794282
- [Background] Rochkind S, Geuna S, Shainberg A. Chapter 25: Phototherapy in peripheral nerve injury: effects on muscle preservation and nerve regeneration. Int Rev Neurobiol. 2009;87:445-64. doi: 10.1016/S0074-7742(09)87025-6. PMID 19682654
- [Background] Oliveira FS, Pinfildi CE, Parizoto NA, Liebano RE, Bossini PS, Garcia EB, Ferreira LM. Effect of low level laser therapy (830 nm) with different therapy regimes on the process of tissue repair in partial lesion calcaneous tendon. Lasers Surg Med. 2009 Apr;41(4):271-6. doi: 10.1002/lsm.20760. PMID 19347936
- [Background] Medeiros DM, Aimi M, Vaz MA, Baroni BM. Effects of low-level laser therapy on hamstring strain injury rehabilitation: A randomized controlled trial. Phys Ther Sport. 2020 Mar;42:124-130. doi: 10.1016/j.ptsp.2020.01.006. Epub 2020 Jan 10. PMID 31991284
- [Background] Lesnak J, Anderson D, Farmer B, Katsavelis D, Grindstaff TL. VALIDITY OF HAND-HELD DYNAMOMETRY IN MEASURING QUADRICEPS STRENGTH AND RATE OF TORQUE DEVELOPMENT. Int J Sports Phys Ther. 2019 Apr;14(2):180-187. PMID 30997270
- [Background] Higashi RH, Toma RL, Tucci HT, Pedroni CR, Ferreira PD, Baldini G, Aveiro MC, Borghi-Silva A, de Oliveira AS, Renno AC. Effects of low-level laser therapy on biceps braquialis muscle fatigue in young women. Photomed Laser Surg. 2013 Dec;31(12):586-94. doi: 10.1089/pho.2012.3388. PMID 24320801
- [Background] Mechanisms of low level light therapy Michael R. Hamblin, Tatiana N Demidova
- [Background] Hamblin, M. R., Ferraresi, C., Huang, Y.-Y., Freitas, L. F. de, & Carroll, J. D. (2018). Low-level light therapy: Photobiomodulation. SPIE Press. ISBN 9781510614154
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Ferraresi C, Huang YY, Hamblin MR. Photobiomodulation in human muscle tissue: an advantage in sports performance? J Biophotonics. 2016 Dec;9(11-12):1273-1299. doi: 10.1002/jbio.201600176. Epub 2016 Nov 22. PMID 27874264
- [Background] Ferraresi C, Hamblin MR, Parizotto NA. Low-level laser (light) therapy (LLLT) on muscle tissue: performance, fatigue and repair benefited by the power of light. Photonics Lasers Med. 2012 Nov 1;1(4):267-286. doi: 10.1515/plm-2012-0032. PMID 23626925
- [Background] Ferraresi C, Bertucci D, Schiavinato J, Reiff R, Araujo A, Panepucci R, Matheucci E Jr, Cunha AF, Arakelian VM, Hamblin MR, Parizotto N, Bagnato V. Effects of Light-Emitting Diode Therapy on Muscle Hypertrophy, Gene Expression, Performance, Damage, and Delayed-Onset Muscle Soreness: Case-control Study with a Pair of Identical Twins. Am J Phys Med Rehabil. 2016 Oct;95(10):746-57. doi: 10.1097/PHM.0000000000000490. PMID 27088469
- [Background] Dos Reis FA, da Silva BA, Laraia EM, de Melo RM, Silva PH, Leal-Junior EC, de Carvalho Pde T. Effects of pre- or post-exercise low-level laser therapy (830 nm) on skeletal muscle fatigue and biochemical markers of recovery in humans: double-blind placebo-controlled trial. Photomed Laser Surg. 2014 Feb;32(2):106-12. doi: 10.1089/pho.2013.3617. Epub 2014 Jan 23. PMID 24456143
- [Background] Dornelles MP, Fritsch CG, Sonda FC, Johnson DS, Leal-Junior ECP, Vaz MA, Baroni BM. Photobiomodulation therapy as a tool to prevent hamstring strain injuries by reducing soccer-induced fatigue on hamstring muscles. Lasers Med Sci. 2019 Aug;34(6):1177-1184. doi: 10.1007/s10103-018-02709-w. Epub 2019 Jan 3. PMID 30607719
- [Background] Cressoni MD, Dib Giusti HH, Casarotto RA, Anaruma CA. The effects of a 785-nm AlGaInP laser on the regeneration of rat anterior tibialis muscle after surgically-induced injury. Photomed Laser Surg. 2008 Oct;26(5):461-6. doi: 10.1089/pho.2007.2150. PMID 18800950
- [Background] Chow RT, Johnson MI, Lopes-Martins RA, Bjordal JM. Efficacy of low-level laser therapy in the management of neck pain: a systematic review and meta-analysis of randomised placebo or active-treatment controlled trials. Lancet. 2009 Dec 5;374(9705):1897-908. doi: 10.1016/S0140-6736(09)61522-1. Epub 2009 Nov 13. PMID 19913903
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Borges LS, Cerqueira MS, dos Santos Rocha JA, Conrado LA, Machado M, Pereira R, Pinto Neto O. Light-emitting diode phototherapy improves muscle recovery after a damaging exercise. Lasers Med Sci. 2014 May;29(3):1139-44. doi: 10.1007/s10103-013-1486-z. Epub 2013 Nov 21. PMID 24258312
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Barbero M, Moresi F, Leoni D, Gatti R, Egloff M, Falla D. Test-retest reliability of pain extent and pain location using a novel method for pain drawing analysis. Eur J Pain. 2015 Sep;19(8):1129-38. doi: 10.1002/ejp.636. Epub 2015 Jan 6. PMID 25565607
- [Background] Bangsbo J, Mohr M, Krustrup P. Physical and metabolic demands of training and match-play in the elite football player. J Sports Sci. 2006 Jul;24(7):665-74. doi: 10.1080/02640410500482529. PMID 16766496
- [Background] Azuma RHE, Merlo JK, Jacinto JL, Borim JM, da Silva RA, Pacagnelli FL, Nunes JP, Ribeiro AS, Aguiar AF. Photobiomodulation Therapy at 808 nm Does Not Improve Biceps Brachii Performance to Exhaustion and Delayed-Onset Muscle Soreness in Young Adult Women: A Randomized, Controlled, Crossover Trial. Front Physiol. 2021 Jun 10;12:664582. doi: 10.3389/fphys.2021.664582. eCollection 2021. PMID 34177615
- [Background] Al-Watban FA, Zhang XY, Andres BL. Low-level laser therapy enhances wound healing in diabetic rats: a comparison of different lasers. Photomed Laser Surg. 2007 Apr;25(2):72-7. doi: 10.1089/pho.2006.1094. PMID 17508840

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT07224646/Prot_SAP_000.pdf